CLINICAL TRIAL: NCT07020507
Title: Exploratory Study to Evaluate the Efficacy of the Cosmetic Product RV3895A on Re-epidermised Scars Following Burns and Surgical Stitches in Adults, Adolescents and Children Over a 6-month Follow-up Period
Status: Terminated | Type: Observational
Why Stopped: Due to recruitment difficulties, the number of subjects included (n=35) was lower than expected (n=60).
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Other Study IDs: RV3895A20210368
Record Dates: First submitted 2025-06-04; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Skin Scars; Post-burn Scars; Post-surgical-stitches Scars

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group 1A: Adults with post-burn scar(s)
  Interventions: Other: Product gel RV3895A
- Group 1C: Adults with post-suture scar(s) requiring stitches to be inserted and removed if applicable (in the case of non-absorbable stitches).
  Interventions: Other: Product gel RV3895A
- Group 2A: Children/adolescents with post-burn scar(s).
  Interventions: Other: Product gel RV3895A

INTERVENTIONS:
Other: Product gel RV3895A — The product is applied twice a day to the scar(s) under study, avoiding all contact with natural orifices (and avoiding ingestion by children in the case of application to the hands in particular). The product is applied using a specific massage technique developed for the product and which is explained by the investigator at visit 1. The product is applied in sufficient quantity to cover the application area.

SUMMARY:
This study is exploratory, non-comparative and open-label, conducted in France. It aims to provide insights into the effectiveness and safety of RV3895A - RY1774, potentially benefiting participants by improving scar appearance and quality of life.The aim of this study is to evaluate the efficacy of the cosmetic product RV3895A - RY1774 on re-epidermised scars of the face and body following burns and surgical stitches in adults, adolescents and children over a 6-month follow-up period.

Patients are divided into 2 groups:

* Group 1: adults with:
* Subgroup 1A: adults with post-burn scar(s)
* Subgroup 1C: adults with post-surgical scar(s) requiring stitches to be inserted and removed if applicable (in the case of non-absorbable stitches).
* Group 2: children and/or adolescents including children aged 2 to 7 years inclusive with:
* Subgroup 2A: children/adolescents with post-burn scar(s)

The study consists of 4 visits:

Visit 1: Inclusion (Day 1), Visit 2: Intermediate visit (Day 22), Visit 3: Intermediate visit (Day 85), Visit 4: End-of-study visit (planned or anticipated) (Day 169 )

ELIGIBILITY:
INCLUSION CRITERIA :

* Male or female
* For group 1: subjects aged between 18 to 65 included
* For group 2: subjects aged between 2 to 17 years included
* Subject with superficial scar(s):

  * Red and re-epidermised
  * Less than 6 months old
  * For subgroups 1A and 2A: Located on the body and/or face
  * For sub-group 1C: Located on the upper limbs and/or neck and/or face
  * For group 1A: spread over an area less than or equal to 30% of the body surface area
  * For group 1C: spread over an area less than or equal to 15% of the body surface area
  * For group 2: spread over an area less than or equal to 10% of the body surface area
  * For sub-groups 1A and 2A: deep 2nd degree burns, whether grafted or not and/or in the 3rd degree graft(s) with limited cutaneous involvement and preservation of underlying structures
  * For sub-group 1C: post-surgical suture requiring stitches to be inserted and removed if applicable (case of non-absorbable stitches)

NON-INCLUSION CRITERIA:

* Subject with abundant hairiness on the instrumental measurement area
* Subject with a known history of scarring problems such as keloid scars
* Subject with superinfected scar(s)
* Subject with non-re-epidermised scar(s)
* Subject with contraindications to scar massage according to investigator assessment (dermatological conditions, treatment, pathologies, etc.) apart from a stage of scarring or a type of scar that does not allow scar massage (e.g. inflammatory scar).
* Subject with another dermatological condition (including pityriasis versicolor, severe pigmentation disorders (vitiligo, melasma, multiple lentigines, numerous and/or congenital nevi in particular if extensive)) or characteristics (e.g. tattoo) on the studied scar(s), liable to interfere with the study evaluations, or considered hazardous for the subject or incompatible with the study requirements, in the opinion of the investigator
* Subject with a pathology that may interfere with the healing stages (such as vascular pathologies, diabetes, chronic smoking associated with vascular complications...)
* Systemic treatments derived from vitamin A (retinoids, etc.) taken within the 2 months before the inclusion visit or planned during the study
* Systemic treatment with corticosteroids and/or immunosuppressants taken within the 4 weeks before the inclusion visit or planned during the study
* Surgery (other than that which caused the scar(s)) or chemical or significantly invasive dermatological treatment on the studied scar(s) liable to interfere, according to investigator assessment, with the study results within the previous weeks before the inclusion visit or planned during the study
* Systemic or topical treatments on the studied scar(s) having an influence on pruritus (benzodiazepines, antihistamines...) established or modified within the weeks before the inclusion visit or planned to be established or modified during the study and considered as not stabilised according to investigator assessment
* Topical corticosteroid and/or immunosuppressants treatments applied on the studied scar(s) within 2 weeks before the inclusion visit or planned during the study
* Silicone-based scar treatment/product(s) applied within the wound healing phase to the studied scar(s)
* Any other scar care product(s) (emollient, etc.) applied on the studied scar(s) within the week before the inclusion visit*
* Water applied on the studied scar(s) within 2 hours before the inclusion * Other medicinal or physical treatments for the scar(s) are authorised (clothing/compressive dressings, massages, stabilised topical antihistamines, thermal water, etc.).

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects were recruited from their usual consultations and/or from the centre's registry. If necessary, advertisements were used.
  Subjects corresponding to the eligibility criteria could receive a telephone call, letter or email offering them to take part in this clinical study.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
Physical aspect of scar(s) compared to normal skin by the investigator | Day 1, Day 22, Day 85, and Day 169
  The investigator assessed the physical appearance of the studied scar(s) in comparison to normal skin using the "POSAS Observer Scale" (Patient and Observer Scar Assessment Scale)
Physical and functional aspect of scar(s) by the subject | Day 1, Day 22, Day 85, and Day 169, and monthly at home between Visit 2 and Visit4
  Subjects who were of age to complete the assessment evaluated the physical appearance in comparison to normal skin and the functional appearance of the studied scar(s) using the "POSAS Patient Scale"
Soothing effect | at Day 1 (before and after product application), Day 22, Day 85, and Day 169, and monthly at home between Visit 2 and Visit 4.
  The subject/parent(s) or legal guardian(s) evaluated the soothing effect using a Numerical Rating Scale (NRS) to assess discomfort over the past 3 days (except for the evaluation at Day 1 after application) from 0 (no discomfort) to 10 (severe discomfort)
Inflammatory aspect of scar | at Day 1, Day 22, Day 85, and Day 169
  The investigator evaluated the inflammatory aspect of the scar using the vitropression test
Evolution of scar aspect compared to Day 1 | at Day 22, Day 85, and Day 169
  The investigator assessed the evolution of the scar's appearance compared to D1 based on all parameters evaluated in the study using a dynamic Investigator's Global Assessment (IGA) scale ranging from -1 (worsening), 0 (no change), 1 (slight improvement), 2 (clear improvement), 3 (very clear improvement)
Overall satisfaction with Test product (Investigator's assessment) | at Day 22, Day 85, and Day 169
  The investigator assessed overall satisfaction with the product's impact on scar appearance based on usual practice and study parameters using an NRS from 0 (not at all satisfied) to 10 (very satisfied)
Overall satisfaction with Test product (Subject/Parent/Guardian assessment) | at Day 22, Day 85, and Day 169
  The subject/parent(s) or legal guardian(s) assessed overall satisfaction with the product's impact on scar appearance using an NRS from 0 (not at all satisfied) to 10 (very satisfied)
Erythema quantification | at Day 1, Day 22, Day 85, and Day 169
  Erythema was quantified using chromametry through spectrocolorimetric parameters
Dermatology Life Quality Index (DLQI) | at Day 1, Day 22, Day 85, and Day 169 and monthly at home between Visit 2 and Visit 4
  Quality of life was assessed by subjects of appropriate age using the Dermatology Life Quality Index (DLQI) questionnaire
Specific impact of burns on quality of life | at Day 1, Day 22, Day 85, and Day 169
  For subgroup 1a (Burns) only : evaluated by subjects using the "body image" and "heat sensitivity" subdomains of the Burn Specific Health Scale-Brief (BSHS-B)
Visual aspect of the scar through illustrative photographs | at Day 1, Day 22, Day 85, and Day 169.
The quantity of product used calculated by weighing the tubes | Between Day 1 and Day 169
Subjective cosmetic acceptability of the product | at Day 22, Day 85, and Day 169
  The subjective cosmetic acceptability of the product was evaluated by the subject/parent(s) or legal guardian(s) using a questionnaire
Recording of adverse events | at Day 1 (first application of the product on site), Day 22, Day 85, and Day 169
  At each visit, the occurrence of adverse events since the last visit was determined based on spontaneous reports from the subject/parent(s) or legal guardian(s), non-subjective questioning, and clinical evaluations performed by the investigator. All adverse events were recorded in the Case Report Form (CRF)
Overall tolerance assessed by the investigator | at Day 22, Day 85, and Day 169
  Overall tolerance was assessed by the investigator considering all individual adverse events and their characteristics, as well as past experience with similar products, using a 5-point scale (Excellent, Very Good, Good, Moderate, Poor)
Compliance | Duration of the study, from Day 1 to Day 169
  The subject was to record in their subject diary the applications of the study product, as well as any omissions and changes in frequency

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique de Rééducation et de Réadaptation Fonctionnelle du Docteur Jean Ster, Lamalou-les-Bains, France